CLINICAL TRIAL: NCT03217929
Title: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) for Food Craving in Obese Individuals: a Randomized, Sham-controlled, Double Blind Clinical Trial.
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) for Food Craving in Obese Individuals.
Acronym: taVNS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ruth Bartelli Grigolon, Master, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 51355115.8.0000.5479
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Obesity; Craving
Keywords: vagus nerve; obesity; craving; food
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-taVNS (Active Comparator)
  Interventions: Device: Active-taVNS
- Sham-taVNS (Sham Comparator)
  Interventions: Device: Sham-taVNS

INTERVENTIONS:
Device: Active-taVNS — Stimulation will be performed using the Neurodyn II (Ibramed) equipment approved by the national regulatory agency (ANVISA). The following parameters will be used: 120 Hz (hertz) of frequency, 250 μs of pulse duration and 12 milliamperes of intensity for a continuous stimulation for 30 minutes. This intensity corresponds to a non-painful mild paresthesia without muscle contraction previously described and evaluated. The 25 cm² (centimeters) electrodes will be positioned over the retroauricular area. A total of 10 sessions (one session per day during 10 week-days) will be performed. Every session will be followed by an interview with a trained psychiatrist to evaluate possible adverse effects and guarantee safety issues regarding the study itself.
  Arms: Active-taVNS
Device: Sham-taVNS — Regarding sham protocol, the device will be turned off after 60 seconds of stimulation without the knowledge of the patient. After this initial period, the referred paresthesia seems to diminish due to nerve accommodation.
  Arms: Sham-taVNS

SUMMARY:
Background: Obesity is one of the most important diseases around the globe; with a continuous increase and public health concern. Current treatments present some limitations. Craving is a symptom usually noticeable and has been described as a "strong desire or urge to use", especially with foods. The vagus nerve and its relations to the neurocircuitry of the reward system play essential roles in food intake regulation and this can be done transcutaneously trough the auricular branch of the vagus nerve (taVNS). Based on the neurobiology of food craving and on the initial data on taVNS demonstrating safety and efficacy in open-label and randomized sham controlled trials, the investigators propose the first randomized, sham controlled, triple-blind trial on taVNS for food craving in obesity.

Methods: This will be a two-arm, triple-blinded, randomized controlled trial with 54 subjects with food craving assigned to either: 1) a 10-session treatment protocol of real taVNS, or 2) a 10-session treatment protocol of sham taVNS, besides qualitative electroencephalogram (qEEG) and heart rate variability (HRV). Participants will be evaluated for primary outcome measures (Food Craving Questionnaire - State [FCQ-S] and Food Craving Questionnaire - Trait [FCQ-T]) before and after intervention, with a follow-up visit of 30 days after the end of treatment. A comparison between sham and active groups will be performed in three occasions [baseline (T1), at the end of the stimulation protocol (T2) and 30 days after the last day of stimulation (T3)].

Discussion: Given the epidemiological situation and economic and social burdens, the possibility of modulating the reward system neurocircuitry trough the vagus nerve with an easy-to-use, low-cost, safe and potential at-home use could represent a breakthrough in treating obesity. The investigators hypothesized that food craving in obese individuals would decrease at least 50%, as well as their intake of high fat, high sugar and processed food, commonly described as palatable foods. Beyond that, the investigators expect that these individuals would improve anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI)>29
* Age between 18 and 55 years old
* Food Craving Questionnaire-State and Trait (FCQ-S and FCQ-T)>108
* Agreement to participate and sign the informed consent term before any procedure is conducted.

Exclusion Criteria:

* History of head injury or epilepsy
* Body metallic implants and pacemaker
* Current use or in the previous six months of psychotropic or anorexigenic medications, recreational drugs and/or participation in weight-loss programs
* Pregnancy or breastfeeding
* Indication of hospitalization
* Substance dependence
* Psychiatric disorder, except for anxiety disorders
* Personality disorders
* Suicidal ideation
* Non-controlled clinical comorbidities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of 40% of food craving symptoms | Baseline, at the end of the stimulation protocol (10 days after) and 30 days after the last day of stimulation.
  Changes in food craving will be evaluated by the Brazilian version of the FCQ-S and FCQ-T. A comparison between sham and active groups will be performed in three occasions.

SECONDARY OUTCOMES:
Decrease of 10% of BMI and hip/waist ratio | Baseline, at the end of the stimulation protocol (10 days after) and 30 days after the last day of stimulation.
Improve metabolic profile. | Baseline, at the end of the stimulation protocol (10 days after) and 30 days after the last day of stimulation.
Improve anxiety symptoms evaluated by the Inventory for Depressive Symptoms (Self-Report version). | Baseline, at the end of the stimulation protocol (10 days after) and 30 days after the last day of stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth B Grigolon, Master, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided